CLINICAL TRIAL: NCT04870320
Title: A Pilot Study of A Novel Cognitive Intervention for Cancer Survivors
Brief Title: Study of Attention and Memory Treatments for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19803; NCI-2021-02024 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Endeavor) (Experimental): Patients play Endeavor over 25 minutes daily 5 days a week for 4 weeks.
  Interventions: Behavioral: Endeavor: Computer-Based Cognitive Stimulation Intervention; Other: Quality of Life (QOL) Questionnaires
- Arm II (Words!) (Active Comparator): Patients play Words! over 25 minutes daily 5 days a week for 4 weeks.
  Interventions: Behavioral: Words!: Computer-Based Cognitive Stimulation Intervention; Other: Quality of Life (QOL) Questionnaires

INTERVENTIONS:
Behavioral: Endeavor: Computer-Based Cognitive Stimulation Intervention — Endeavor application will be utilized by participant on iPad
  Other Names: Computer-Based Cognitive Stimulation Intervention; Computer-Based General Cognitive Stimulation Intervention
  Arms: Arm I (Endeavor)
Behavioral: Words!: Computer-Based Cognitive Stimulation Intervention — Words! application will be utilized by participant on iPad
  Other Names: Computer-Based Cognitive Stimulation Intervention; Computer-Based General Cognitive Stimulation Intervention
  Arms: Arm II (Words!)
Other: Quality of Life (QOL) Questionnaires — Standardized QOL questionnaire will be administered at each study visit

SUMMARY:
This clinical trial investigates if certain electronic games may be effective in improving attention and memory function in cancer survivors. Cancer related cognitive impairment (CRCI) is an issue experienced by many cancer patients/survivors. CRCI includes perceived or objective problems with memory, executive function, and attention/concentration. CRCI has a negative impact on survivors' ability to work, carry out routine activities, and engage in social and family relationships. CRCI may result in significant distress and reduced quality of life. Certain electronic games may help improve attention and memory function in cancer survivors and reduce symptoms of CRCI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the recruitment and retention rates for both arms of this study. II. Determine the effect size for changes in cognitive function (i.e., Test of Variables of Attention (TOVA) [i.e. attention], Adaptive Cognitive Evaluation (ACE) [i.e. working memory]) in the intervention group compared to the control group following the 4-week study.

III. Evaluate adherence rates for and satisfaction with the interventions. IV. Evaluate for treatment-related adverse events (e.g., nausea, motion sickness).

SECONDARY OBJECTIVE:

I. To determine effect sizes for depression, fatigue, and sleep disturbance, by comparing changes in the intervention group to changes in the control group, following the 4-week study.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients play Endeavor over 25 minutes daily 5 days a week for 4 weeks.

ARM II: Patients play Words! over 25 minutes daily 5 days a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Attention Function Index (AFI) score of < 7.5
* Are able to read, write, and understand English
* Ability to understand an electronic informed consent document, and the willingness to sign it
* Have a Karnofsky performance status (KPS) score of >= 50
* Have access to WiFi connection

Exclusion Criteria:

* Receiving active treatment for cancer recurrence
* Have significant cognitive impairment
* Have sensory or motor deficits that prevent them from doing the assessment and using the application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who completed the study | Up to 6 weeks
  Completion is defined as participants who completed all 4 weeks of intervention and final assessment.
Mean change in scores on the Test of Variables of Attention (TOVA) over time | Up to 4 weeks
  The TOVA records responses to visual or auditory stimuli through the participants iPAD, with a unique, highly accurate +/1 millisecond (ms) microswitch. The TOVA (Copyright 1991- 2021 by The TOVA Company) automatically calculates response time variability (consistency), response time (speed), commissions (impulsivity), and omissions (focus and vigilance). Results are reported as standard scores (average = 100 with a standard deviation of 15) and are compared to a large normative sample stratified by gender and age. Scores above 85 are within normal limits, 80-85 are borderline, and below 80 are not within normal limits. The mean change in scores will be estimated as the norm-based standardized difference in means from enrollment (Week 1) to the last assessment (Week 4).
Percent change in scores on the TOVA over time | Up to 4 weeks
  The TOVA records responses to visual or auditory stimuli through the participants iPAD, with a unique, highly accurate +/1 millisecond (ms) microswitch. The TOVA (Copyright 1991- 2021 by The TOVA Company) automatically calculates response time variability (consistency), response time (speed), commissions (impulsivity), and omissions (focus and vigilance). Results are reported as standard scores (average = 100 with a standard deviation of 15) and are compared to a large normative sample stratified by gender and age. Scores above 85 are within normal limits, 80-85 are borderline, and below 80 are not within normal limits. Will be estimated as the standardized difference between the groups in the percent score change from enrollment (Week 1) to the last assessment (Week 4).
Mean changes in Adaptive Cognitive Evaluation (ACE) | Up to 4 weeks
  The ACE is a mobile cognitive control assessment battery containing standard tests that assess different aspects of cognitive control (attention, working memory, and goal management), modified by incorporating adaptive algorithms, immersive graphics, video tutorials, motivating feedback, and a user-friendly interface. The ACE is administered to all participants via iPad and the scores will be estimated as the standardized difference in means from enrollment (Week 1) to the last assessment (Week 4).
Percent change in scores on the ACE over time | Up to 4 weeks
  The ACE is a mobile cognitive control assessment battery containing standard tests that assess different aspects of cognitive control (attention, working memory, and goal management), modified by incorporating adaptive algorithms, immersive graphics, video tutorials, motivating feedback, and a user-friendly interface. The ACE is administered to all participants via iPad and the scores will be estimated as the standardized difference between the groups in the percent score change from enrollment (Week 1) to the last assessment (Week 4).
Proportion of time using application | Up to 4 weeks
  Adherence rate will be evaluated by comparing the amount of time the participant should have used the application to the actual amount of time the participant used the application.
Percentage of participants who experienced treatment-related adverse events | Up to 6 weeks
  Safety analyses will involve examination of and comparison between groups for the percentage of participants by adverse event severity and type of treatment-related adverse events. Comparisons of the frequencies between groups will be conducted using Chi-square or Fisher's exact test.

SECONDARY OUTCOMES:
Change in mean severity scores on the Center for Epidemiologic Studies - Depression Scale (CES-D) | Up to 4 weeks
  The CES-D scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past week. Responses are rated on a 5 point Likert scale with response option ranging 0="Rarely or none of the time (less than 1 day )" to 4='Most or all of the time (5-7 days)". The scoring of positive items is reversed. Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology and will be estimated as the standardized difference in means of each measure at the last assessment from enrollment to the last assessment.
Change in mean severity scores on the Lee Fatigue Scale | Up to 4 weeks
  The Lee Fatigue Scale is used to measure the impact of fatigue on a participants quality of life. The scale consists of 18 items relating to the subjective experience of fatigue. Each item is rated on a 0 to 10 numeric rating scale (e.g., from "not at all tired" to "extremely tired"). Scores can range from 0 to 10. The instrument has two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10). The fatigue subscale score is calculated as the mean of the 13 fatigue items and the energy subscale score is the mean of the 5 energy items. Higher scores on the fatigue subscale represent greater fatigue severity, and higher scores on the energy subscale indicate higher levels of energy and will be estimated as the standardized difference in means of each measure at the last assessment from enrollment to the last assessment.
Change in severity scores on the General Sleep Disturbance Scale (GSDS) | Up to 4 weeks
  The GSDS consists of 21 items related to frequency in the past month of difficulty getting to sleep when respondents were asked to think about the past month, and each response is on a 8-point Likert scale from 0 ("never") to 7 ("all the time"). Will be estimated as the standardized difference in means of each measure at the last assessment, and as the difference between the groups in the percent change from enrollment to the last assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Miaskowski, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No